CLINICAL TRIAL: NCT00632216
Title: Multicenter and Prospective Study to Determine the Satisfaction With Actonel (Risedronate Sodium) 35mg Once a Week Using Biochemical Markers of Bone as a Control, in Postmenopausal Women With Osteoporosis
Brief Title: A Study to Determine the Satisfaction With Actonel in Postmenopausal Women With Osteoporosis
Acronym: ROSPA-CTx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: YEU Wang/Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISED_L_01054
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Risedronate Sodium

SUMMARY:
The study in the labeled and real conditions of prescription of Actonel will investigate the satisfaction of patients with its new formulation: 35 mg Once A Week. The study will also measure response rates in CTX (the C-telopeptide of type I collagen) at baseline and after 12 weeks of treatment with risedronate 35 mg Once A Week.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal outpatients women > 55 and < 70 years who have a clinical presentation appropriate for treatment of established osteoporosis based on the investigator's clinical judgment (a T-score for BMD (DEXA) of lumbar spine or femoral neck less than or equal to - 2.5 from an assessment performed at screening or within 12 months prior to the screening visit or evidence of previous vertebral fracture).

Exclusion Criteria:

* History of Cancer: Basal Cell or Squamous Cell carcinoma-documented 6-month remission.
* Diagnosis of hypocalcemia, hyperparathyroidism, hyperthyroidism.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2004-05; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To determine the satisfaction of subject with Actonel 35 mg | Once a Week in the treatment of postmenopausal osteoporosis

SECONDARY OUTCOMES:
To measure response rates in CTX with Actonel 35 mg | Once A Week

CONTACTS AND LOCATIONS:
Overall Officials: YEU Wang, Study Director — Sanofi